CLINICAL TRIAL: NCT04016558
Title: Evaluating Affective and Unified Behavioral Approaches to Reducing Diabetes Distress and Improving Glycemic Control
Brief Title: Behavioral Approaches to Reducing Diabetes Distress and Improving Glycemic Control
Acronym: EMBARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 133107A; R01DK121241-02 (NIH)
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes; Diabetes Distress
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- StreamLine (Experimental): Diabetes education, behavioral management
  Interventions: Behavioral: StreamLine
- TunedIn (Experimental): Diabetes distress reduction, emotion regulation techniques.
  Interventions: Behavioral: TunedIn
- FixIt (Experimental): Unified program combining diabetes education, behavioral management, diabetes distress reduction, and emotion regulation techniques.
  Interventions: Behavioral: FixIt

INTERVENTIONS:
Behavioral: StreamLine — StreamLine is an education/disease management program that focuses on systematic methods to identify and resolve specific blood glucose problems, primarily through changes in carbohydrate consumption, and use of basal and bolus insulin. Participants will attend a brief, four-hour meeting with a Certified Diabetes Educator (CDE) and, using standardized blood glucose data, will learn how to employ a five-point blood glucose management system to identify and resolve blood glucose problems (e.g., excursions, lows) that have the greatest HbA1c or hypoglycemic impacts.
  Participants will then meet individually (30 minutes) with their CDE to review their blood glucose data, identify a specific blood glucose problem, and use the five-point program to create a plan to address the problem. Four additional individual meetings (30 minutes) will occur at approximately two to three-week intervals to best support individualized and participant-tailored management-change efforts.
  Arms: StreamLine
Behavioral: TunedIn — TunedIn utilizes emotion regulation-based strategies to help participants observe that how they feel affects what they do regarding diabetes management. Participants will attend two highly interactive group workshops (6 hours followed by 2 hours) facilitated by a psychologist or social worker experienced in diabetes. Each will identify and discuss common emotional responses related to blood glucose management (e.g., over-reacting, avoiding, and lack of mindfulness).
  Between the two workshops (two weeks), participants will complete a "feeling log" to document feelings, situation/context, and resolution around specific management events. Two individual meetings with the interventionist (30 minutes) will allow participants to identify and address a specific diabetes distress-related problem. Four web-based video group meetings (60 minutes, monthly) will continue to support participants over time.
  Arms: TunedIn
Behavioral: FixIt — FixIt combines components of StreamLine and TunedIn to allow participants to explore feelings and expectations alongside the identification of problematic blood glucose patterns. StreamLine will be co-facilitated by a psychologist/social worker experienced in diabetes and a CDE. Participants will attend two group workshops (six hours followed by four hours), separated by two weeks.
  Between the two workshops, participants will record their blood glucose data and keep a parallel "feeling log" to provide context. Four individual meetings with an interventionist (30 minutes) will allow participants to identify and address a specific blood glucose problem and create a plan to address it. Full discussion of diabetes distress-related aspects of the plan will take place to enhance mindfulness and identify typical emotion regulation strategies to ease problem resolution. Three web-based video group meetings (60 minutes, monthly) will continue to support participants over time.
  Arms: FixIt

SUMMARY:
This study is comparing three programs to reduce Diabetes Distress (the worries and concerns that people with diabetes may experience as they struggle to keep blood glucose levels in range) in adults with type 1 diabetes. About a third of participants will take part in the TunedIn program, about a third will take part in the FixIt program, and about a third in the StreamLine program.

DETAILED DESCRIPTION:
Diabetes Distress (DD) is the personal, often hidden side of diabetes: it reflects the unique emotional burdens and strains that individuals with diabetes may experience as they struggle to keep blood glucose levels within range. When high, DD can have a major, negative impact on disease management and glycemic control. High DD is characterized by frustration, feeling overwhelmed, and feeling hopeless and discouraged by the unceasing demands of diabetes. DD is also linked to an individual's beliefs, expectations, current life situation, and personal and social resources.

The proposed study is a three-arm, 12-month randomized comparison trial to test the added value of a DD-targeted (TunedIn) intervention vs. a unified DD and management intervention (FixIt), relative to a traditional, educational/behavioral-management intervention (StreamLine). Each of the three programs (arms) will follow a separate, standardized protocol. All participants will receive three months of intervention with nine months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with type 1 diabetes (confirmed by clinical history and/or anti-glutamic acid decarboxylase] antibody testing) on intensive insulin treatment;
* Diagnosis of type 1 diabetes for at least 12 months that occurred at or below age 40;
* Have a recent HbA1c of 7.5% or higher;
* Not have started to use any new (to the participant) diabetes device (such as an insulin pump or continuous glucose monitor) in the past 6 months;
* Internet access through a computer or smart phone;
* Ability to speak/read English.

Exclusion Criteria:

* No documented psychosis, blindness, dementia, active dialysis, substance abuse, amputations, or severe functional deficits, or recent major surgery or hospitalization in the past year.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Hessler, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher L, Hessler D, Polonsky WH, Masharani U, Guzman S, Bowyer V, Strycker L, Ahmann A, Basina M, Blumer I, Chloe C, Kim S, Peters AL, Shumway M, Weihs K, Wu P. T1-REDEEM: A Randomized Controlled Trial to Reduce Diabetes Distress Among Adults With Type 1 Diabetes. Diabetes Care. 2018 Sep;41(9):1862-1869. doi: 10.2337/dc18-0391. Epub 2018 Jul 5. PMID 29976567
- [Background] Fisher L, Hessler D, Polonsky W, Strycker L, Guzman S, Bowyer V, Blumer I, Masharani U. Emotion regulation contributes to the development of diabetes distress among adults with type 1 diabetes. Patient Educ Couns. 2018 Jan;101(1):124-131. doi: 10.1016/j.pec.2017.06.036. Epub 2017 Jul 8. PMID 28739179
- [Background] Hessler DM, Fisher L, Polonsky WH, Masharani U, Strycker LA, Peters AL, Blumer I, Bowyer V. Diabetes distress is linked with worsening diabetes management over time in adults with Type 1 diabetes. Diabet Med. 2017 Sep;34(9):1228-1234. doi: 10.1111/dme.13381. Epub 2017 Jun 18. PMID 28498610
- [Background] Fisher L, Hessler D, Polonsky W, Strycker L, Masharani U, Peters A. Diabetes distress in adults with type 1 diabetes: Prevalence, incidence and change over time. J Diabetes Complications. 2016 Aug;30(6):1123-8. doi: 10.1016/j.jdiacomp.2016.03.032. Epub 2016 Apr 4. PMID 27118163
- [Background] Fisher L, Polonsky WH, Hessler DM, Masharani U, Blumer I, Peters AL, Strycker LA, Bowyer V. Understanding the sources of diabetes distress in adults with type 1 diabetes. J Diabetes Complications. 2015 May-Jun;29(4):572-7. doi: 10.1016/j.jdiacomp.2015.01.012. Epub 2015 Feb 7. PMID 25765489

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred virtually (email and phone contact)
Groups:
- StreamLine: Diabetes education, behavioral management
  StreamLine: StreamLine is an education/disease management program that focuses on systematic methods to identify and resolve specific blood glucose problems, primarily through changes in carbohydrate consumption, and use of basal and bolus insulin. Participants will attend a brief, four-hour meeting with a Certified Diabetes Educator (CDE) and, using standardized blood glucose data, will learn how to employ a five-point blood glucose management system to identify and resolve blood glucose problems (e.g., excursions, lows) that have the greatest HbA1c or hypoglycemic impacts.
  Participants will then meet individually (30 minutes) with their CDE to review their blood glucose data, identify a specific blood glucose problem, and use the five-point program to create a plan to address the problem. Four additional individual meetings (30 minutes) will occur at approximately two to three-week intervals to best support individualized and participant-tailored management-change efforts.
- TunedIn: Diabetes distress reduction, emotion regulation techniques.
  TunedIn: TunedIn utilizes emotion regulation-based strategies to help participants observe that how they feel affects what they do regarding diabetes management. Participants will attend two highly interactive group workshops (6 hours followed by 2 hours) facilitated by a psychologist or social worker experienced in diabetes. Each will identify and discuss common emotional responses related to blood glucose management (e.g., over-reacting, avoiding, and lack of mindfulness).
  Between the two workshops (two weeks), participants will complete a "feeling log" to document feelings, situation/context, and resolution around specific management events. Two individual meetings with the interventionist (30 minutes) will allow participants to identify and address a specific diabetes distress-related problem. Four web-based video group meetings (60 minutes, monthly) will continue to support participants over time.
- FixIt: Unified program combining diabetes education, behavioral management, diabetes distress reduction, and emotion regulation techniques.
  FixIt: FixIt combines components of StreamLine and TunedIn to allow participants to explore feelings and expectations alongside the identification of problematic blood glucose patterns. StreamLine will be co-facilitated by a psychologist/social worker experienced in diabetes and a CDE. Participants will attend two group workshops (six hours followed by four hours), separated by two weeks.
  Between the two workshops, participants will record their blood glucose data and keep a parallel "feeling log" to provide context. Four individual meetings with an interventionist (30 minutes) will allow participants to identify and address a specific blood glucose problem and create a plan to address it. Full discussion of diabetes distress-related aspects of the plan will take place to enhance mindfulness and identify typical emotion regulation strategies to ease problem resolution. Three web-based video group meetings (60 minutes, monthly) will continue to support participants over time.
Period: Overall Study
Arm/Group | StreamLine | TunedIn | FixIt
Started | 101 | 97 | 98
Received Intervention | 97 | 91 | 88
Completed | 89 | 77 | 78
Not Completed | 12 | 20 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | StreamLine | TunedIn | FixIt | Total
Number analyzed (Participants) | 101 | 97 | 98 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (15.2) | 47.6 (15.3) | 42.5 (15.4) | 46.3 (15.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 23 | 18 | 17 | 58
  Gender: Female | 77 | 76 | 80 | 233
  Gender: Female to male (transgender) | 1 | 2 | 0 | 3
  Gender: Male to female (transgender) | 0 | 1 | 0 | 1
  Gender: Unknown | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 9 | 33
  Not Hispanic or Latino | 87 | 82 | 88 | 257
  Unknown or Not Reported | 2 | 3 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 5 | 8
  White | 89 | 89 | 86 | 264
  More than one race | 5 | 5 | 4 | 14
  Unknown or Not Reported | 3 | 1 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 101 | 97 | 98 | 296
T1-DDS (total diabetes distress) mean score [Mean (Standard Deviation); unit: units on a scale] — Diabetes distress is measured on a 1-6 scale and calculated as a mean score. A higher score indicates more distress.
  units on a scale | 2.8 (0.8) | 2.8 (0.8) | 3.0 (0.7) | 2.8 (0.8)
HbA1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 8.2 (0.8) | 8.2 (0.9) | 8.4 (1.1) | 8.3 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Diabetes Distress at 12 Months
Description: Self-reported diabetes distress across several domains will be assessed using the Type 1 Diabetes Distress Scale (T1-DDS) a validated measure averaged across items (range 1.0-6.0 with higher scores indicating a higher level of diabetes-related distress).
Time Frame: 12 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | StreamLine | TunedIn | FixIt
Number analyzed (Participants) | 97 | 91 | 88
score on a scale | 2.34 (0.074) | 2.03 (0.077) | 2.06 (0.079)
Statistical Analysis 1: Comparison: StreamLine vs TunedIn vs FixIt; Test type: Superiority; p = .007, ANCOVA; Mean Difference (Final Values) = 0.28

2. Primary Outcome: Hemoglobin A1c (HbA1c) at 12 Months
Description: Hemoglobin A1c (HbA1c) assay laboratory result
Time Frame: 12 months
Measure: Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | StreamLine | TunedIn | FixIt
Number analyzed (Participants) | 97 | 91 | 88
percentage of glycosylated hemoglobin | 7.52 (0.092) | 7.60 (0.098) | 7.94 (0.101)
Statistical Analysis 1: Comparison: StreamLine vs TunedIn vs FixIt; Test type: Superiority; p = .006, ANCOVA; Mean Difference (Final Values) = 0.42

3. Secondary Outcome: Hypoglycemic Episodes at 12 Months
Description: Self-reported number of severe of hypoglycemic episodes in the past 6 months, or since the last assessment. A numeric count is reported, zero indicates no hypoglycemic episodes, and a higher number indicates more hypoglycemic episodes.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: hypoglycemic episodes
Arm/Group | StreamLine | TunedIn | FixIt
Number analyzed (Participants) | 97 | 91 | 88
hypoglycemic episodes | 1.17 (1.15) | 1.32 (1.66) | 1.23 (1.46)
Statistical Analysis 1: Comparison: StreamLine vs TunedIn vs FixIt; Test type: Superiority; p = 0.82, ANCOVA; Mean Difference (Final Values) = 0.15

4. Secondary Outcome: Depression Symptoms at 12 Months
Description: Symptoms of depression will be measured using the self-completion Patient Health Questionnaire (PHQ-8). The score ranges from zero to 24 with a higher score indicating more symptoms of depression.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | StreamLine | TunedIn | FixIt
Number analyzed (Participants) | 97 | 91 | 88
score on a scale | 6.35 (5.72) | 5.94 (4.54) | 7.09 (5.73)
Statistical Analysis 1: Comparison: StreamLine vs TunedIn vs FixIt; Test type: Superiority; p = .01, ANCOVA; Mean Difference (Final Values) = 1.15

5. Secondary Outcome: Missed Insulin Boluses at 12 Months
Description: Self-reported number of missed or skipped insulin boluses in the past week
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of insulin boluses skipped
Arm/Group | StreamLine | TunedIn | FixIt
Number analyzed (Participants) | 97 | 91 | 88
percentage of insulin boluses skipped | 0.15 (0.15) | 0.17 (0.16) | 0.19 (0.17)
Statistical Analysis 1: Comparison: StreamLine vs TunedIn vs FixIt; Test type: Superiority; p = .40, ANCOVA; Mean Difference (Final Values) = 0.04

6. Secondary Outcome: Nonreactivity to Inner Experience at 12 Months
Description: Nonreactivity to inner experience will be assessed by the nonreactivity sub-scale of the Five Facet Mindfulness Questionnaire. Items are scored from 1-5 with items summed to calculate a total scale score. The total score ranges from 7-35. Higher scores indicate greater nonreactivity to inner emotional experiences.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | StreamLine | TunedIn | FixIt
Number analyzed (Participants) | 97 | 91 | 88
score on a scale | 23.68 (5.29) | 24.34 (5.18) | 24.22 (5.00)

7. Secondary Outcome: Non-judging of Experience at 12 Months
Description: Non-judging of experience will be assessed by the nonjudgmental subscale of the Five Facet Mindfulness Questionnaire. Individual items are scored on a 1-5 scale and then summed to calculate a scale score with higher scores indicating greater non-judging of emotional experience. The total score ranges from 8-40.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | StreamLine | TunedIn | FixIt
Number analyzed (Participants) | 97 | 91 | 88
score on a scale | 31.29 (7.55) | 32.13 (5.90) | 30.48 (6.99)
Statistical Analysis 1: Comparison: StreamLine vs TunedIn vs FixIt; Test type: Superiority; p = .12, ANCOVA; Mean Difference (Final Values) = 1.65

8. Secondary Outcome: Personal Control Over Illness at 12 Months
Description: The personal control subscale from the Revised Illness Perception Questionnaire will assess participants' perceived control over their illness. The items are scored on a 1-5 scale and summed across items for a total score with higher scores indicating greater personal control. The total score ranges from 6-30.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | StreamLine | TunedIn | FixIt
Number analyzed (Participants) | 97 | 91 | 88
score on a scale | 24.77 (3.23) | 24.68 (2.70) | 24.99 (2.97)
Statistical Analysis 1: Comparison: StreamLine vs TunedIn vs FixIt; Test type: Superiority; p = .39, ANCOVA; Mean Difference (Final Values) = 0.22

9. Secondary Outcome: Self-compassion - Diabetes (SCS-D) at 12 Months
Description: Diabetes-specific self-compassion will be measured using the validate Self-Compassion Scale - Diabetes (SCS-D) in which the average of items is calculated. Items are scored on a scale from 1 to 5 with higher scores indicative of greater self compassion.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | StreamLine | TunedIn | FixIt
Number analyzed (Participants) | 97 | 91 | 88
score on a scale | 3.42 (0.85) | 3.60 (0.81) | 3.44 (0.94)
Statistical Analysis 1: Comparison: StreamLine vs TunedIn vs FixIt; Test type: Superiority; p < .01, ANCOVA; Mean Difference (Final Values) = 0.18

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of consent/baseline to 12 month follow-up.
Arm/Group | StreamLine | TunedIn | FixIt
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/91 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/91 | 0/88
Other Adverse Events (participants affected / at risk) | 0/97 | 0/91 | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT04016558/Prot_SAP_000.pdf